CLINICAL TRIAL: NCT02019732
Title: Burden of Mild Outcomes Due to Influenza in the United States, July 2000 Through April 2009 and October 2010 to May 2011
Brief Title: Study to Assess the Burden of Mild Outcomes (Physician Office Visits) Due to Influenza in the United States
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 117233
Record Dates: First submitted 2013-11-27; First posted 2013-12-24 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Influenza
Keywords: Mild outcomes; Database; Influenza-attributable; Retrospective; Influenza; United States of America (USA)
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Study Group: Applicable subjects less than 65 years of age identified in the Marketscan Commercial database during the period from July 2000 through April 2009, and October 2010 to May 2011 and subjects 65 years of age and older identified in MarketScan Medicare Supplemental database during the period from July 2006 through April 2009, and October 2010 to May 2011.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection from existing electronic healthcare databases (Marketscan Commercial database, MarketScan Medicare Supplemental database).

SUMMARY:
This is a database study to quantify the burden of multiple mild outcomes (i.e., those that result in visits to a physician's office) attributable to influenza in the United States, stratified by age group, geographic region and influenza subtype for selected influenza seasons.

DETAILED DESCRIPTION:
This is a retrospective database study to quantify the burden of multiple mild pre-defined influenza-attributable outcomes of interest, which resulted in physician office visits for persons who were less than 65 years of age, in the United States in the relevant Marketscan Commercial database in the period from July 2000 through April 2009, and October 2010 to May 2011. The corresponding physician office visits for persons 65 years of age and older, with a mild influenza-attributable outcome of interest, in the United States that were recorded in the relevant MarketScan Medicare Supplemental database in the period from July 2006 through April 2009, and October 2010 to May 2011 were also investigated. The period from April 2009 through September 2010 is excluded to avoid the H1N1 pandemic wave.

ELIGIBILITY:
Inclusion Criteria:

• Recorded in a Marketscan database with any of the specified diagnostic codes.

Exclusion Criteria:

• Missing data in any of the following fields: age, diagnosis, region or visit date.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All records related to physician office visits of subjects less than 65 years of age and 65 years of age and older in the United States with an outcome of interest in the relevant Marketscan database.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Weekly occurrences of potentially influenza-attributable physician's office visits by age, region and season. | Up to 10 years approximately (Marketscan Commercial Database) and up to 6 years approximately (Marketscan Medicare Supplemental Database).
  - All the events contained within "potentially influenza-attributable" office visits. - Weekly proportion of circulating influenza A and B strains determined for each season.

SECONDARY OUTCOMES:
Assessment of Influenza vaccine content and effectiveness by season. | Up to 10 years approximately (Marketscan Commercial Database) and up to 6 years approximately (Marketscan Medicare Supplemental Database).
Assessment of Influenza vaccine coverage by season and region. | Up to 10 years approximately (Marketscan Commercial Database) and up to 6 years approximately (Marketscan Medicare Supplemental Database).
Assessment of Influenza B vaccine mismatch (by region and season). | Up to 10 years approximately (Marketscan Commercial Database) and up to 6 years approximately (Marketscan Medicare Supplemental Database).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Matias G, Haguinet F, Lustig RL, Edelman L, Chowell G, Taylor RJ. Model estimates of the burden of outpatient visits attributable to influenza in the United States. BMC Infect Dis. 2016 Nov 7;16(1):641. doi: 10.1186/s12879-016-1939-7. PMID 27821091